CLINICAL TRIAL: NCT01355211
Title: Diagnostic Utility of Emergency Electroencephalography in Identifying Non-convulsive Seizure and Subclinical Status Epilepticus in Patients With Altered Mental Status
Brief Title: Putting Electroencephalography (EEG) in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Bio-Signal Group Corp. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); State University of New York - Downstate Medical Center (Other); Kings County Hospital Department of Emergency Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RC3NS070658 (NIH); RC3NS070658 (NIH)
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Altered Mental Status; Generalized Nonconvulsive Seizure Disorder; Status-epilepticus
Keywords: Altered Mental Status; non-convulsive seizure; status epilepticus; electroencephalography
MeSH Terms: conditions — Epilepsy, Generalized; Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the proposed research is to compare the diagnostic accuracy of a portable wireless electroencephalography (EEG) device (Biosignal Micro-EEG) to standard EEG in identifying abnormal EEG patterns (mainly non-convulsive seizure and non-convulsive status epilepticus) in emergency department (ED) patients with altered mental status. Comparing the the accuracy of EEG recordings and interpretations of Micro-EEG to those of standard EEG will allow the investigators to assess the utility of this novel device in the ED patients with altered mental status. The unique qualities of Micro-EEG device could potentially facilitate easier access to EEG test in all ED patients.

This study will also provide valid information regarding the prevalence of non-convulsive seizure in ED patients with altered mental status.The gold standard for diagnosing non-convulsive seizure would be standard EEG.

All study participants will undergo electroencephalography using the two devices (standard EEG and micro-EEG) and a combination of standard electrodes and Electro-Cap in a randomized order: 1. Standard EEG with standard EEG electrodes, 2. Micro-EEG with standard EEG electrodes, and 3. Micro-EEG with Electro-Cap electrodes.

DETAILED DESCRIPTION:
Formulated Research Question:

Population: ED patients with altered mental status (AMS) Intervention: Micro-EEG Comparison: Standard EEG Outcomes: 1. Sensitivity, specificity, positive/negative likelihood ratios of micro-EEG in identifying non-convulsive seizures and abnormal brain activities 2. The concordance of EEG interpretations between micro-EEG and standard EEGs recordings Design Prospective cross-sectional

Definitions:

Altered Mental Status: Any acute change in level of arousability or responsiveness (e.g. confusion, lethargy, delirium, coma, aphasia, disinhibition, labile/blunted affect or unexpected psychosis).

Types of AMS (for the purpose of the study):

1. AMS alone
2. AMS with non-specific motor activity (subtle motor movement such as eye blinking, nystagmus, focal motor movements, or myoclonus)
3. Prolonged AMS following one or more tonic-clonic seizures suggesting status epilepticus Non-convulsive seizure (NCZ):A seizure without clonic or tonic activity or other convulsive motor activity.

Status Epilepticus (SE):SE is defined as 1. More than 30 minutes of continuous seizure activity or 2. Two or more sequential seizures without recovery of consciousness between seizures.

ELIGIBILITY:
Inclusion Criteria:

ED patients ≥ 13 year-old with AMS on arrival to ED

Exclusion Criteria:

1. Patients with apparent and immediately correctable cause of AMS upon presentation (determined by ED attending physician during initial evaluation):

   * Patients with finger stick or serum glucose less than 60 mg/dl
   * Patients with hypothermia
   * Patients with hyperthermia, heat exhaustion or heat stroke
   * Patients with opioid overdose responding to Narcan
2. Patients who cannot undergo EEG recordings because of severe head and injury, hemodynamic instability, transfer to operating room, etc.)
3. Hemodynamically unstable patients (SBP < 90 mmHg)
4. Uncooperative or combative patients on whom the EEG simply cannot be obtained.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 260 patients will be recruited for the study. Adult and pediatric patients ≥ 13 year-old with AMS on arrival to ED
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic Utility of Emergency Electroencephalography in Identifying Non-convulsive Seizure and Subclinical Status Epilepticus in Patients with Altered Mental Status (AMS) | 6 months
  1. Sensitivity, specificity, positive/negative likelihood ratios of micro-EEG in identifying non-convulsive seizures and abnormal brain activities
  2. The concordance of EEG interpretations between micro-EEG and standard EEG recordings

CONTACTS AND LOCATIONS:
Overall Officials: Shahriar Zehtabchi, MD, Principal Investigator — Recruiting
Locations (1):
- 450 Clarkson Avenue, Brooklyn, New York, United States

REFERENCES:
- [Derived] Zehtabchi S, Abdel Baki SG, Omurtag A, Sinert R, Chari G, Malhotra S, Weedon J, Fenton AA, Grant AC. Prevalence of non-convulsive seizure and other electroencephalographic abnormalities in ED patients with altered mental status. Am J Emerg Med. 2013 Nov;31(11):1578-82. doi: 10.1016/j.ajem.2013.08.002. Epub 2013 Sep 23. PMID 24070982